CLINICAL TRIAL: NCT02710968
Title: Study of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in Fetuses With Severe Left Congenital Diaphragmatic Hernia (CDH)
Brief Title: Fetoscopic Endoluminal Tracheal Occlusion (FETO) for Severe Left Diaphragmatic Hernia (CDH)
Acronym: FETO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00054901
Record Dates: First submitted 2015-08-17; First posted 2016-03-17 (Estimated); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: FETO
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 11540KE and Balt Goldbal 2 balloon (Experimental): Patients meeting inclusion criteria will receive fetoscopic tracheal occlusion using the fetoscopy sheath 11540 KE and the Balt Goldbal2 detachable balloon.
  Participants with an O/E LHR <25% (severe group) will have FETO completed at 27 weeks + 0 days to 29 weeks + 6 days gestation. Balloon removal is 4-5 weeks after that.
  Participants with an O/E LHR 25 to <30% (less severe group) will have FETO completed at 30 weeks + 0 days to 31 weeks + 6 days gestation. Balloon removal is 3 - 4 weeks after that.
  Interventions: Device: 11540KE and Balt Goldbal 2 balloon

INTERVENTIONS:
Device: 11540KE and Balt Goldbal 2 balloon — Fetoscopic tracheal occlusion will be performed using above devices and reversed after 4-5 weeks.
  Other Names: Karl Storz 11540 KE fetoscopy sheath; BALT GOLDBAL2 1.5 mm detachable balloon; BALT COAX delivery catheter (BALTACCIBDPE100)

SUMMARY:
Despite advances in prenatal diagnosis and postnatal therapies, including extracorporeal membrane oxygenation (ECMO), inhaled nitric oxide therapy, and ventilator strategies that minimize ventilator-induced lung injury, morbidity and mortality rates for babies with congenital diaphragmatic hernia (CDH) remain high. The survival relates to the degree of prenatal lung compression and the subsequent impairment of pulmonary function following delivery. Prenatal assessment by ultrasound or magnetic resonance imaging allows to estimate the severity by relating the circumference of the lung contralateral to the hernia to the fetal head circumference lung to head ratio (LHR) and by noting the degree of upward herniation of the liver. Based on the observed to expected lung to head ratio (O/E LHR), prenatally diagnosed congenital diaphragmatic hernia can be prognostically assessed. While overall survival of congenital diaphragmatic hernia is approximately 60%, an O/E LHR <25% is associated with survival between 11-24%.

The rationale for fetal therapy in severe congenital diaphragmatic hernia is to restore adequate lung growth for neonatal survival. Prenatal tracheal occlusion obstructs the normal egress of lung fluid during pulmonary development leading to increased lung tissue stretch, increased cell proliferation, and accelerated lung growth. European colleagues have developed intrauterine endoscopic techniques (fetoscopy) to position and remove endoluminal tracheal balloons in utero (fetoscopic endotracheal occlusion = FETO). Recently, the Belgium group published summary results of FETO showing an improved survival in 175 patients with isolated left CDH from 24% to 49%. We hypothesize that FETO can be performed and may increase survival and decrease morbidity when compared to standard prenatal care for the treatment of severe CDH in the most severe group of fetuses with left CDH (O/E LHR < 30%). FETO therapy will be considered in two subgroups: those with and O/E LHR <25% (severe group) and those with an O/E between 25 to <30% (less severe group).

DETAILED DESCRIPTION:
Comprehensive fetal evaluations will be completed at the Johns Hopkins Center for Fetal Therapy to confirm eligibility. This includes an ultrasound, magnetic resonance imaging, a fetal echocardiogram and fetal genetic studies to identify cases with isolated CDH. Participant must be willing to remain under supervision of the Center for Fetal Therapy at the Johns Hopkins Hospital while the fetal airway is occluded.

Participants will undergo FETO with standardized preoperative, intraoperative, post-operative care, and delivery. The FETO will be timed between 27+0 to 29+6 weeks gestation for fetuses with an O/E LHR <25% and between 30+0 to 31+6 weeks gestation for fetuses with an O/E LHR between 25% to <30%. Fetal analgesia and immobilization will consist of fentanyl, atropine and vecuronium. A 10 Fr cannula, 1.3 mm fetoscope within a 3.3 mm sheath (Karl Storz, Tuttlingen, Germany), and a detachable balloon occlusion (BALTACCI-BDPE, Balt, Montmorency, France) system will be used.

Serial ultrasound measurements of lung volume and LHR will begin within 24-48 hours following surgery and continue weekly. Amniotic fluid level and membrane status will also be monitored at weekly intervals. Ultrasonography for fetal growth will be performed every 4 weeks.

All discharged participants and their support person need to remain within 30 minutes of the surgery center until delivery to permit standardized postoperative management. The social worker at the Center for Fetal Therapy will serve as the participant advocate and assist families in identifying subsidized appropriate accommodation as required. Participants will be on modified bed rest for the first 2 weeks post discharge, but subsequently allowed to graduate to moderate activity if the uterus is quiescent.

At 34+0 weeks to 34 + 6 weeks, participants will undergo removal of the tracheal balloon. Balloon retrieval can be either by in utero puncture by ultrasound-guided percutaneous needling or fetoscopic retrieval. In the event there is a need for emergent balloon removal prior to 34 weeks due to the development of preterm labor, shortening of the cervix, preterm rupture of membranes, abnormally vigorous lung response, or development of fetal hydrops, delivery by EXIT or cesarean section will be performed. If percutaneous puncture of balloon is unsuccessful prior to delivery, immediate bronchoscopy and establishment of airway will be performed. Maternal corticosteroids (betamethasone 12 mg intramuscularly and repeated once at 24 hours) will be administered 48 hours prior to fetoscopic balloon removal (due to risks of preterm delivery associated with instrumentation) or for impending preterm delivery.

Timing for induction of labor at 37 weeks to 39 weeks will depend upon favorable status of the cervix. Cesarean section will be based upon standard obstetrical indications. In regards to postnatal care, a resuscitation team from neonatology and pediatric surgery will be present at delivery. A standardized protocol will be utilized for postnatal care, using lung protection strategy.

Continued follow-up of children until age 2 is planned as the current standard of care. These follow-ups may include bronchoscopy, brain imaging, audiology exam, pulmonary function testing, chest radiograph and developmental assessment.

The study duration per mother and child will be up to 877 days, with up to 82 days screening, up to 55 days in the intervention phase, and 744 days in delivery and follow-up.

Follow-up will be conducted from birth to 24 months of age at which time the study will conclude.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years and older, who are able to consent.
* Singleton pregnancy.
* Anatomically and chromosomally normal fetus.
* Left sided diaphragmatic hernia with liver up.
* SEVERE pulmonary hypoplasia with O/E LHR < 30%.
* In patients with O/E LHR 25% to <30%, enrollment prior to gestational age 30 weeks+0 days to 31 weeks+6 days.
* In patients with O/E LHR <25%, enrollment prior to gestational age 27 weeks+0 days to 29 weeks+6 days.

Exclusion Criteria:

* Pregnant women < 18 years.
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy.
* Technical limitations precluding fetoscopic surgery.
* Women with history of natural rubber latex allergy.
* Preterm labor, cervix shortened <15 mm within 24 hours prior to the FETO balloon insertion or uterine anomaly strongly predisposing to preterm labor, placenta previa.
* Diaphragmatic hernia: right-sided or bilateral, major associated anomalies, isolated left-sided with the O/E LHR ≥ 30%.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Successful balloon insertion and removal | 4 to 7 weeks
  The feasibility of performing the procedure, managing the pregnancy during the period of tracheal occlusion, and removal of the device prior to delivery at Johns Hopkins Hospital.

SECONDARY OUTCOMES:
Survival | 28 days after delivery
  The neonatal survival of participants receiving FETO expressed as a percentage of the total number of participants undergoing the procedure.
Percentage of lung growth | 4 to 7 weeks
  The percentage of size increase in the contralateral fetal lung as related to the pre-procedure lung size

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet A Baschat, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Fetal Therapy, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Claus F, Sandaite I, DeKoninck P, Moreno O, Cruz Martinez R, Van Mieghem T, Gucciardo L, Richter J, Michielsen K, Decraene J, Devlieger R, Gratacos E, Deprest JA. Prenatal anatomical imaging in fetuses with congenital diaphragmatic hernia. Fetal Diagn Ther. 2011;29(1):88-100. doi: 10.1159/000320605. Epub 2010 Nov 9. PMID 21063073
- [Background] Danzer E, Gerdes M, Bernbaum J, D'Agostino J, Bebbington MW, Siegle J, Hoffman C, Rintoul NE, Flake AW, Adzick NS, Hedrick HL. Neurodevelopmental outcome of infants with congenital diaphragmatic hernia prospectively enrolled in an interdisciplinary follow-up program. J Pediatr Surg. 2010 Sep;45(9):1759-66. doi: 10.1016/j.jpedsurg.2010.03.011. PMID 20850617
- [Background] Deprest JA, Hyett JA, Flake AW, Nicolaides K, Gratacos E. Current controversies in prenatal diagnosis 4: Should fetal surgery be done in all cases of severe diaphragmatic hernia? Prenat Diagn. 2009 Jan;29(1):15-9. doi: 10.1002/pd.2108. No abstract available. PMID 19125386
- [Background] Luks FI, Deprest JA, Vandenberghe K, Laermans I, De Simpelaere L, Brosens IA, Lerut T. Fetoscopy-guided fetal endoscopy in a sheep model. J Am Coll Surg. 1994 Jun;178(6):609-12. PMID 8193755
- [Background] Deprest J, Nicolaides K, Done' E, Lewi P, Barki G, Largen E, DeKoninck P, Sandaite I, Ville Y, Benachi A, Jani J, Amat-Roldan I, Gratacos E. Technical aspects of fetal endoscopic tracheal occlusion for congenital diaphragmatic hernia. J Pediatr Surg. 2011 Jan;46(1):22-32. doi: 10.1016/j.jpedsurg.2010.10.008. PMID 21238635
- [Background] Harrison MR, Adzick NS, Flake AW, VanderWall KJ, Bealer JF, Howell LJ, Farrell JA, Filly RA, Rosen MA, Sola A, Goldberg JD. Correction of congenital diaphragmatic hernia in utero VIII: Response of the hypoplastic lung to tracheal occlusion. J Pediatr Surg. 1996 Oct;31(10):1339-48. doi: 10.1016/s0022-3468(96)90824-6. PMID 8906657
- [Background] Benachi A, Chailley-Heu B, Delezoide AL, Dommergues M, Brunelle F, Dumez Y, Bourbon JR. Lung growth and maturation after tracheal occlusion in diaphragmatic hernia. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):921-7. doi: 10.1164/ajrccm.157.3.9611023. PMID 9517613
- [Background] De Paepe ME, Johnson BD, Papadakis K, Sueishi K, Luks FI. Temporal pattern of accelerated lung growth after tracheal occlusion in the fetal rabbit. Am J Pathol. 1998 Jan;152(1):179-90. PMID 9422535
- [Background] Bratu I, Flageole H, Laberge JM, Chen MF, Piedboeuf B. Pulmonary structural maturation and pulmonary artery remodeling after reversible fetal ovine tracheal occlusion in diaphragmatic hernia. J Pediatr Surg. 2001 May;36(5):739-44. doi: 10.1053/jpsu.2001.22950. PMID 11329579
- [Background] Davey MG, Hedrick HL, Bouchard S, Mendoza JM, Schwarz U, Adzick NS, Flake AW. Temporary tracheal occlusion in fetal sheep with lung hypoplasia does not improve postnatal lung function. J Appl Physiol (1985). 2003 Mar;94(3):1054-62. doi: 10.1152/japplphysiol.00733.2002. PMID 12571135
- [Background] Bratu I, Flageole H, Laberge JM, Possmayer F, Harbottle R, Kay S, Khalife S, Piedboeuf B. Surfactant levels after reversible tracheal occlusion and prenatal steroids in experimental diaphragmatic hernia. J Pediatr Surg. 2001 Jan;36(1):122-7. doi: 10.1053/jpsu.2001.20027. PMID 11150450
- [Background] Flageole H, Evrard VA, Piedboeuf B, Laberge JM, Lerut TE, Deprest JA. The plug-unplug sequence: an important step to achieve type II pneumocyte maturation in the fetal lamb model. J Pediatr Surg. 1998 Feb;33(2):299-303. doi: 10.1016/s0022-3468(98)90451-1. PMID 9498406
- [Background] Wilson JM, DiFiore JW, Peters CA. Experimental fetal tracheal ligation prevents the pulmonary hypoplasia associated with fetal nephrectomy: possible application for congenital diaphragmatic hernia. J Pediatr Surg. 1993 Nov;28(11):1433-9; discussion 1439-40. doi: 10.1016/0022-3468(93)90426-l. PMID 8301455
- [Background] DiFiore JW, Fauza DO, Slavin R, Peters CA, Fackler JC, Wilson JM. Experimental fetal tracheal ligation reverses the structural and physiological effects of pulmonary hypoplasia in congenital diaphragmatic hernia. J Pediatr Surg. 1994 Feb;29(2):248-56; discussion 256-7. doi: 10.1016/0022-3468(94)90328-x. PMID 8176601
- [Background] Papadakis K, De Paepe ME, Tackett LD, Piasecki GJ, Luks FI. Temporary tracheal occlusion causes catch-up lung maturation in a fetal model of diaphragmatic hernia. J Pediatr Surg. 1998 Jul;33(7):1030-7. doi: 10.1016/s0022-3468(98)90526-7. PMID 9694089
- [Background] Wild YK, Piasecki GJ, De Paepe ME, Luks FI. Short-term tracheal occlusion in fetal lambs with diaphragmatic hernia improves lung function, even in the absence of lung growth. J Pediatr Surg. 2000 May;35(5):775-9. doi: 10.1053/jpsu.2000.6067. PMID 10813348
- [Background] Luks FI, Wild YK, Piasecki GJ, De Paepe ME. Short-term tracheal occlusion corrects pulmonary vascular anomalies in the fetal lamb with diaphragmatic hernia. Surgery. 2000 Aug;128(2):266-72. doi: 10.1067/msy.2000.107373. PMID 10923003
- [Background] Schnitzer JJ, Hedrick HL, Pacheco BA, Losty PD, Ryan DP, Doody DP, Donahoe PK. Prenatal glucocorticoid therapy reverses pulmonary immaturity in congenital diaphragmatic hernia in fetal sheep. Ann Surg. 1996 Oct;224(4):430-7; discussion 437-9. doi: 10.1097/00000658-199610000-00002. PMID 8857848
- [Background] Hedrick HL, Kaban JM, Pacheco BA, Losty PD, Doody DP, Ryan DP, Manganaro TF, Donahoe PK, Schnitzer JJ. Prenatal glucocorticoids improve pulmonary morphometrics in fetal sheep with congenital diaphragmatic hernia. J Pediatr Surg. 1997 Feb;32(2):217-21; discussion 221-2. doi: 10.1016/s0022-3468(97)90182-2. PMID 9044125
- [Background] Schnitzer JJ, Thompson JE, Hedrick HL. A new ventilator improves CO2 removal in newborn lambs with congenital diaphragmatic hernia. Crit Care Med. 1999 Jan;27(1):109-12. doi: 10.1097/00003246-199901000-00037. PMID 9934903
- [Background] Sylvester KG, Rasanen J, Kitano Y, Flake AW, Crombleholme TM, Adzick NS. Tracheal occlusion reverses the high impedance to flow in the fetal pulmonary circulation and normalizes its physiological response to oxygen at full term. J Pediatr Surg. 1998 Jul;33(7):1071-4; discussion 1074-5. doi: 10.1016/s0022-3468(98)90533-4. PMID 9694096
- [Background] Quinn TM, Sylvester KG, Kitano Y, Kitano Y, Liechty KW, Jarrett BP, Adzick NS, Flake AW. TGF-beta2 is increased after fetal tracheal occlusion. J Pediatr Surg. 1999 May;34(5):701-4; discussion 704-5. doi: 10.1016/s0022-3468(99)90359-7. PMID 10359167
- [Background] Kitano Y, Flake AW, Quinn TM, Kanai M, Davies P, Sablich TJ, Schneider C, Adzick NS, von Allmen D. Lung growth induced by tracheal occlusion in the sheep is augmented by airway pressurization. J Pediatr Surg. 2000 Feb;35(2):216-21; discussion 221-2. doi: 10.1016/s0022-3468(00)90012-5. PMID 10693668
- [Background] Davey MG, Danzer E, Schwarz U, Adzick NS, Flake AW, Hedrick HL. Prenatal glucocorticoids and exogenous surfactant therapy improve respiratory function in lambs with severe diaphragmatic hernia following fetal tracheal occlusion. Pediatr Res. 2006 Aug;60(2):131-5. doi: 10.1203/01.pdr.0000227509.94069.ae. PMID 16864691
- [Background] Davey M, Shegu S, Danzer E, Ruchelli E, Adzick S, Flake A, Hedrick HL. Pulmonary arteriole muscularization in lambs with diaphragmatic hernia after combined tracheal occlusion/glucocorticoid therapy. Am J Obstet Gynecol. 2007 Oct;197(4):381.e1-7. doi: 10.1016/j.ajog.2007.06.061. PMID 17904968
- [Background] Dekoninck P, Gratacos E, Van Mieghem T, Richter J, Lewi P, Ancel AM, Allegaert K, Nicolaides K, Deprest J. Results of fetal endoscopic tracheal occlusion for congenital diaphragmatic hernia and the set up of the randomized controlled TOTAL trial. Early Hum Dev. 2011 Sep;87(9):619-24. doi: 10.1016/j.earlhumdev.2011.08.001. PMID 21907109
- [Background] Khan PA, Cloutier M, Piedboeuf B. Tracheal occlusion: a review of obstructing fetal lungs to make them grow and mature. Am J Med Genet C Semin Med Genet. 2007 May 15;145C(2):125-38. doi: 10.1002/ajmg.c.30127. PMID 17436297
- [Background] Flageole H, Evrard VA, Vandenberghe K, Lerut TE, Deprest JA. Tracheoscopic endotracheal occlusion in the ovine model: technique and pulmonary effects. J Pediatr Surg. 1997 Sep;32(9):1328-31. doi: 10.1016/s0022-3468(97)90314-6. PMID 9314255
- [Background] Fayoux P, Marciniak B, Devisme L, Storme L. Prenatal and early postnatal morphogenesis and growth of human laryngotracheal structures. J Anat. 2008 Aug;213(2):86-92. doi: 10.1111/j.1469-7580.2008.00935.x. PMID 19172727
- [Background] Chiba T, Albanese CT, Farmer DL, Dowd CF, Filly RA, Machin GA, Harrison M. Balloon tracheal occlusion for congenital diaphragmatic hernia: experimental studies. J Pediatr Surg. 2000 Nov;35(11):1566-70. doi: 10.1053/jpsu.2000.18311. PMID 11083424
- [Background] Cannie MM, Jani JC, De Keyzer F, Allegaert K, Dymarkowski S, Deprest J. Evidence and patterns in lung response after fetal tracheal occlusion: clinical controlled study. Radiology. 2009 Aug;252(2):526-33. doi: 10.1148/radiol.2522081955. Epub 2009 Jun 9. PMID 19508989
- [Result] Deprest J, Gratacos E, Nicolaides KH; FETO Task Group. Fetoscopic tracheal occlusion (FETO) for severe congenital diaphragmatic hernia: evolution of a technique and preliminary results. Ultrasound Obstet Gynecol. 2004 Aug;24(2):121-6. doi: 10.1002/uog.1711. PMID 15287047
- [Result] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Result] Flake AW, Crombleholme TM, Johnson MP, Howell LJ, Adzick NS. Treatment of severe congenital diaphragmatic hernia by fetal tracheal occlusion: clinical experience with fifteen cases. Am J Obstet Gynecol. 2000 Nov;183(5):1059-66. doi: 10.1067/mob.2000.108871. PMID 11084541
- [Result] Harrison MR, Mychaliska GB, Albanese CT, Jennings RW, Farrell JA, Hawgood S, Sandberg P, Levine AH, Lobo E, Filly RA. Correction of congenital diaphragmatic hernia in utero IX: fetuses with poor prognosis (liver herniation and low lung-to-head ratio) can be saved by fetoscopic temporary tracheal occlusion. J Pediatr Surg. 1998 Jul;33(7):1017-22; discussion 1022-3. doi: 10.1016/s0022-3468(98)90524-3. PMID 9694087
- [Result] Harrison MR, Sydorak RM, Farrell JA, Kitterman JA, Filly RA, Albanese CT. Fetoscopic temporary tracheal occlusion for congenital diaphragmatic hernia: prelude to a randomized, controlled trial. J Pediatr Surg. 2003 Jul;38(7):1012-20. doi: 10.1016/s0022-3468(03)00182-9. PMID 12861529
- [Result] Harrison MR, Keller RL, Hawgood SB, Kitterman JA, Sandberg PL, Farmer DL, Lee H, Filly RA, Farrell JA, Albanese CT. A randomized trial of fetal endoscopic tracheal occlusion for severe fetal congenital diaphragmatic hernia. N Engl J Med. 2003 Nov 13;349(20):1916-24. doi: 10.1056/NEJMoa035005. PMID 14614166
- [Result] Hedrick MH, Estes JM, Sullivan KM, Bealer JF, Kitterman JA, Flake AW, Adzick NS, Harrison MR. Plug the lung until it grows (PLUG): a new method to treat congenital diaphragmatic hernia in utero. J Pediatr Surg. 1994 May;29(5):612-7. doi: 10.1016/0022-3468(94)90724-2. PMID 8035268
- [Result] Schnitzer JJ, Thompson JE, Hedrick HL, Kaban JM, Wilson JM. High-frequency intratracheal pulmonary ventilation: improved gas exchange at lower airway pressures. J Pediatr Surg. 1997 Feb;32(2):203-6. doi: 10.1016/s0022-3468(97)90179-2. PMID 9044122
- [Result] Jani JC, Nicolaides KH, Gratacos E, Vandecruys H, Deprest JA; FETO Task Group. Fetal lung-to-head ratio in the prediction of survival in severe left-sided diaphragmatic hernia treated by fetal endoscopic tracheal occlusion (FETO). Am J Obstet Gynecol. 2006 Dec;195(6):1646-50. doi: 10.1016/j.ajog.2006.04.004. Epub 2006 Jun 12. PMID 16769018
- [Result] Kays DW, Langham MR Jr, Ledbetter DJ, Talbert JL. Detrimental effects of standard medical therapy in congenital diaphragmatic hernia. Ann Surg. 1999 Sep;230(3):340-8; discussion 348-51. doi: 10.1097/00000658-199909000-00007. PMID 10493481
- [Result] Deprest JA, Evrard VA, Verbeken EK, Perales AJ, Delaere PR, Lerut TE, Flageole H. Tracheal side effects of endoscopic balloon tracheal occlusion in the fetal lamb model. Eur J Obstet Gynecol Reprod Biol. 2000 Sep;92(1):119-26. doi: 10.1016/s0301-2115(00)00435-8. PMID 10986445
- [Result] Gallot D, Boda C, Ughetto S, Perthus I, Robert-Gnansia E, Francannet C, Laurichesse-Delmas H, Jani J, Coste K, Deprest J, Labbe A, Sapin V, Lemery D. Prenatal detection and outcome of congenital diaphragmatic hernia: a French registry-based study. Ultrasound Obstet Gynecol. 2007 Mar;29(3):276-83. doi: 10.1002/uog.3863. PMID 17177265
- [Result] Jani J, Nicolaides KH, Keller RL, Benachi A, Peralta CF, Favre R, Moreno O, Tibboel D, Lipitz S, Eggink A, Vaast P, Allegaert K, Harrison M, Deprest J; Antenatal-CDH-Registry Group. Observed to expected lung area to head circumference ratio in the prediction of survival in fetuses with isolated diaphragmatic hernia. Ultrasound Obstet Gynecol. 2007 Jul;30(1):67-71. doi: 10.1002/uog.4052. PMID 17587219
- [Derived] Baschat AA, Rosner M, Millard SE, Murphy JD, Blakemore KJ, Keiser AM, Kearney J, Bullard J, Nogee LM, Bembea M, Jelin EB, Miller JL. Single-Center Outcome of Fetoscopic Tracheal Balloon Occlusion for Severe Congenital Diaphragmatic Hernia. Obstet Gynecol. 2020 Mar;135(3):511-521. doi: 10.1097/AOG.0000000000003692. PMID 32028493